CLINICAL TRIAL: NCT05615467
Title: An Open-Label Study in Healthy Participants to Evaluate the Effect of LY3556050 on Metformin Pharmacokinetics
Brief Title: A Study of Effect of LY3556050 on Metformin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18629; J2P-MC-LXBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-11-11; First posted 2022-11-14 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3556050 + Metformin + Iohexol (Experimental): LY3556050 administered orally in combination with metformin given orally and iohexol given intravenously (IV).
  Interventions: Drug: LY3556050; Drug: Metformin; Drug: Iohexol

INTERVENTIONS:
Drug: LY3556050 — Administered orally.
Drug: Metformin — Administered orally.
Drug: Iohexol — Administered IV.

SUMMARY:
The main purpose of this study is to evaluate how much Metformin gets into the bloodstream and how long the body takes to get rid of it when it is administered orally in combination with LY3556050 in healthy participants. Iohexol will be administered to evaluate kidney function. Each enrolled participant will remain in the study for up to 7 weeks including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation
* Participants with body weight of at least 50 kilograms (kg) or more and have a body mass index (BMI) between 18.5 and 35.0 kilograms per meter squared (kg/m²)
* Have an ECG at screening considered to be within acceptable limits by the investigator
* Male participants who agree to use contraception and female participants of child bearing potential who agree to use contraception and women not of child bearing potential may participate.

Exclusion Criteria:

* Women who are lactating
* Have known allergies or contraindications to LY3556050, metformin, iodine, iohexol, or other contrast agents, related compounds or any components of their formulation, or history of significant atopy
* Have a history, or ECG findings, of clinically significant bradycardia, heart block, tachycardia, sick sinus syndrome/sinoatrial block, first-degree AV block, or second- or third-degree AV block, bundle branch block or other tachy- or brady-arrhythmias; o rhave any other abnormality in the 12-lead ECG that, in the opinion of the investigator, confounds assessment of QT interval or increases the risks associated with participating in the study
* Have active or a history of gastritis or peptic ulcer disease

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Metformin | Predose on day 1 through 13 days postdose
  PK: AUC of Metformin
PK: Maximum Observed Drug Concentration (Cmax) of Metformin | Predose on day 1 through 13 days postdose
  PK: Cmax of Metformin

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PRA International, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No